CLINICAL TRIAL: NCT02804971
Title: Cardiovascular Comorbidities, Inflammation, Aging and Bronchiectasis
Brief Title: Cardiovascular Comorbidities and Bronchiectasis
Acronym: BRONCOCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Principal Investigator, Bernard MAITRE, Pr, Centre Hospitalier Intercommunal Creteil
Other Study IDs: BRONCOCA
Record Dates: First submitted 2016-06-15; First posted 2016-06-17 (Estimated); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Bronchiectasis have multiple etiologies but share a similar bronchial injury associated with inflammation, which leads to a progressive lung deterioration. This disease is responsible for a frequent access to care with an exacerbation rate of 1.8 per year with a high risk of hospitalization. Natural history is marked by recurrent infectious diseases which are the main prognosis factor. This disease is associated with an inflammation rate in the lung as well as in the blood. Up to now, no study has been described comorbidities associated with this chronic disease but our hypothesis is that cardiovascular diseases will be more frequent in these patients. In fact systemic inflammation driven by bronchial infections may increase frequency of cardiovascular diseases.

The investigators decide to conduct a monocentric observational study to define the prevalence and characterization of cardiovascular comorbidities as well as markers of accelerated aging. We would like to test the hypothesis that cardiovascular comorbidities are frequent in bronchiectasis and may be associated with markers of inflammation and aging.

Phenotype of the lung disease will include: spirometry, plethysmography, DLCO measurement according to the ATS/ERS guideline. 6M walking test and echocardiography will be also performed.

Frequency of comorbidities will be calculated with data from questionnaire as well as standardized explorations.

Aging related manifestations will be measured: arterial stiffness using aortic pulse wave velocity, bone mineral density using dual energy X-ray absorptiometry. Appendicular skeletal muscle mass and grip test were also performed.

Blood test were also performed to measure inflammatory markers, cytokines and length of telomere in circulating leucocytes.

DETAILED DESCRIPTION:
Phenotype of the lung disease will include: spirometry, plethysmography, DLCO measurement according to the ATS/ERS guideline. 6M walking test and echocardiography will be also performed.

Frequency of comorbidities will be calculated with data from questionnaire as well as standardized explorations.

Aging related manifestations will be measured: arterial stiffness using aortic pulse wave velocity, bone mineral density using dual energy X-ray absorptiometry. Appendicular skeletal muscle mass and grip test were also performed.

Blood test were also performed to measure inflammatory markers, cytokines and length of telomere in circulating leucocytes.

ELIGIBILITY:
Inclusion Criteria:

* 40 ≤ Age ≤ 80 years
* Formal diagnosis of bronchiectasis by imaging (CT-scan)
* For women, pregnancy test negative
* Affiliation to a social Security
* written inform consent

Exclusion Criteria:

* Patients with a diagnosis of Cystic Fibrosis
* Contre indication of one of the tests
* Exacerbation with hospitalization or outpatient clinic visit in the last 4 weeks.
* Unability to obtain an informed consent
* Pregnancy or Breast feeding

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of bronchiectasis based on imaging in a recent (less than 2 years) CT-scan.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10-25 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of the cardiovascular comorbidities | Examinations / tests required for this primary outcome measure will be performed within the month following the inclusion visit.

SECONDARY OUTCOMES:
Frequency of aging-related abnormalities (higher aortic pulse-wave velocity, lower bone mineral density, lower squelettal muscle mass index) and shorter telomere length in patients. | Examinations / tests required for this secondary outcome measure will be performed within the month following the inclusion visit.
Correlation between the severity of the disease (BSI score) and cardiovascular comorbidities. | Examinations / tests required for this secondary outcome measure will be performed within the month following the inclusion visit.
Correlation between biological markers of aging and inflammation. | Examinations / tests required for this secondary outcome measure will be performed within the month following the inclusion visit.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard MAITRE, Principal Investigator — CHI Créteil
Locations (1):
- Chi Creteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No